CLINICAL TRIAL: NCT03809429
Title: A Randomised, Controlled, Open Label, Parallel Group, Multicentre Trial Comparing the Efficacy and Safety of Individualised FE 999049 (Follitropin Delta) Dosing, Using a Long GnRH Agonist Protocol and a GnRH Antagonist Protocol in Women Undergoing Controlled Ovarian Stimulation
Brief Title: Follitropin Delta in Long GnRH Agonist and GnRH Antagonist Protocols (BEYOND)
Acronym: BEYOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000304; 2017-002783-40 (EudraCT Number)
Record Dates: First submitted 2019-01-07; First posted 2019-01-18 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2022-09

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — FE 999049; Gonadotropin-Releasing Hormone; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FE 999049 + GnRH agonist (GONAPEPTYL) (Experimental)
  Interventions: Drug: FE 999049 + GnRH agonist (GONAPEPTYL)
- FE 999049 + GnRH antagonist (CETROTIDE) (Active Comparator)
  Interventions: Drug: FE 999049 + GnRH antagonist (CETROTIDE)

INTERVENTIONS:
Drug: FE 999049 + GnRH agonist (GONAPEPTYL) — Pre-filled injection pen
  Arms: FE 999049 + GnRH agonist (GONAPEPTYL)
Drug: FE 999049 + GnRH antagonist (CETROTIDE) — Powder and solvent for solution for injection
  Arms: FE 999049 + GnRH antagonist (CETROTIDE)

SUMMARY:
To compare the efficacy and safety of FE 999049 (follitropin delta) and its personalized dosing algorithm in controlled ovarian stimulation for in vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI) using a long gonadotropin-releasing hormone (GnRH) agonist protocol versus a short GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women aged 18-40 undergoing their first IVF/ICSI cycle that are in good physical and mental health and that have been diagnosed with problems in the fallopian tubes, mild endometriosis or have partners with decreased sperm quality.
* The participants must have a regular menstrual cycle, a normal uterus and 2 normal ovaries.
* The allowed body mass index is 17.5-32 Kg/m^2.

Exclusion Criteria:

* Women with very high ovarian reserve, strong preference for either treatment, severe endometriosis, history of repeated miscarriage, couples with known problems in the chromosomes, history or high risk of producing blood cloths, women known to have chronic diseases, women recently participating in trials with non-registered drugs.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing their first IVF/ICSI cycle and aged 18-40 years will be included.
Enrollment: 437 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (16):
- Austria (3):
  - Das Kinderwunsch Institut Schenk GmbH, Dobl
  - Kepler University Hospital Linz, Linz
  - Kinderwunschzentrum Goldenes Kreuz Privatklinik, Vienna
- Rigshospitalet, Copenhagen, Denmark
- Israel (4):
  - Hillel Yafe Medical Center, Hadera
  - Shaare Zedek Medical Center, Jerusalem
  - Beilinson Hospital Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Dipartimento della Donna, del bambino e delle malattie urologiche, Bologna
  - European Hospital, Roma
- Netherlands (2):
  - St. Elisabeth Ziekenhuis, Tilburg
  - Isala Fertility Center, Zwolle
- Norway (3):
  - Oslo University Hospital, Oslo
  - Sykehuset Telemark HF, Porsgrunn
  - Medicus AS, Trondheim
- Gyn-A.R.T. AG, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lobo R, Soerdal T, Ekerhovd E, Cohlen B, Porcu E, Schenk M, Shufaro Y, Smeenk J, Suerdieck MB, Pinton P, Pinborg A; BEYOND Investigators. BEYOND: a randomized controlled trial comparing efficacy and safety of individualized follitropin delta dosing in a GnRH agonist versus antagonist protocol during the first ovarian stimulation cycle. Hum Reprod. 2024 May 9;39(7):1481-94. doi: 10.1093/humrep/deae092. Online ahead of print. PMID 38723189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was opened for recruitment in April 2019, and participants were assessed at 16 investigational sites in 7 countries between May 2019 and Feb 2022.
Pre-assignment Details: In total, 532 participants were screened of which 437 were randomized. Of the 437 participants, 435 participants were included in the Full Analysis Set (FAS): 220 participants to long GnRH agonist and 215 participants to GnRH antagonist. 406 participants were exposed to the investigational medicinal product (IMP): 202 participants to long GnRH agonist and 204 participants to GnRH antagonist.
  Two participants discontinued before the start of stimulation with FE999049 due to COVID-19 pandemic.
Period: Overall Study
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Started (The number covers the number of randomized participants.) | 220 | 215
Completed | 192 | 195
Not Completed | 28 | 20
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Adverse Event | 6 | 9
Not completed — COVID-19 | 3 | 1
Not completed — Participant was discontinued by investigator | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE) | Total
Number analyzed (Participants) | 220 | 215 | 435
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (4.4) | 32.4 (4.2) | 32.3 (4.3)
Age, Customized [Count of Participants; unit: Participants]
  <35 years | 143 | 141 | 284
  35-37 years | 47 | 48 | 95
  38-40 years | 30 | 26 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 215 | 435
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 211 | 205 | 416
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  White | 208 | 202 | 410
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 29 | 31 | 60
  Netherlands | 31 | 26 | 57
  Norway | 117 | 114 | 231
  Denmark | 15 | 16 | 31
  Italy | 9 | 12 | 21
  Israel | 13 | 12 | 25
  Switzerland | 6 | 4 | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.36 (3.50) | 24.39 (3.55) | 24.37 (3.52)

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Description: The number of oocytes retrieved was recorded at the oocyte retrieval visit.
Time Frame: On day of oocyte retrieval (up to 22 days after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Oocytes
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Oocytes | 11.1 (5.9) | 9.6 (5.5)
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Test type: Other; p = 0.0185, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = 1.31, 95% CI 2-sided [0.22 to 2.40]

2. Secondary Outcome: Proportion of Subjects With Cycle Cancellation Due to Poor Ovarian Response or Excessive Ovarian Response
Description: For each participant, the reason for cycle cancellation was recorded
Time Frame: At end-of-stimulation (up to 20 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
participants
  Excessive response | 2 | 3
  Poor response | 1 | 3
  Other reason | 1 | 1

3. Secondary Outcome: Proportion of Subjects With Blastocyst Transfer Cancellation After Oocyte Retrieval Due to (Risk of) Ovarian Hyperstimulation Syndrome (OHSS)
Description: For each participant, the reason for blastocyst transfer cancellation was recorded.
Time Frame: At end of transfer (up to 4 weeks)
Population: Participants analyzed for this endpoint represent participants with blastocyst transfer cancellation.
Measure: Number; unit: participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 27 | 30
participants
  Transfer cancellation | 27 | 30
  Reason for transfer cancellation: Adverse Event | 5 | 8
  Reason for transfer cancellation: Risk of OHSS | 1 | 1
  Reason for transfer cancellation: No blastocyst | 13 | 18
  Reason for transfer cancellation: COVID-19 | 3 | 1
  Reason for transfer cancellation: Other reason | 5 | 2

4. Secondary Outcome: Number of Follicles
Description: The total number of follicles and the number of follicles per size category will be reported
Time Frame: On stimulation day 6 and at end-of-stimulation (up to 20 days)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Number of follicles
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Number of follicles
  Total number of follicles at Stimulation Day 6 | 15.2 (6.3) | 14.9 (6.3)
  Follicles >= 10 mm at Stimulation Day 6 | 4.6 (4.3) | 7.1 (3.6)
  Follicles >= 12 mm at Stimulation Day 6 | 1.6 (2.7) | 3.8 (2.9)
  Total number of follicles at End-of-stimulation visit | 18.3 (7.1) | 17.1 (8.0)
  Follicles >= 10 mm at End-of-stimulation visit | 14.8 (6.4) | 13.3 (6.1)
  Follicles >= 12 mm at End-of-stimulation visit | 12.2 (5.3) | 10.9 (5.1)
  Follicles >= 15 mm at End-of-stimulation visit | 7.9 (3.7) | 7.2 (3.3)
  Follicles >= 17 mm at End-of-stimulation visit | 4.8 (2.1) | 4.6 (2.0)
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); >=10 mm at end of stimulation; Test type: Other; p = 0.0281, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = 1.14, 95% CI 2-sided [0.12 to 2.15]
Statistical Analysis 2: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); >=12 mm at end of stimulation; Test type: Other; p = 0.0258, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = 0.99, 95% CI 2-sided [0.12 to 1.86]
Statistical Analysis 3: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); >=15 mm at end of stimulation; Test type: Other; p = 0.0672, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = 0.58, 95% CI 2-sided [-0.04 to 1.20]
Statistical Analysis 4: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); >=17 mm at end of stimulation; Test type: Other; p = 0.3390, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = 0.21, 95% CI 2-sided [-0.22 to 0.63]

5. Secondary Outcome: Proportion of Subjects With <4, 4-7, 8-14, 15-19 and ≥20 Oocytes Retrieved
Description: Grouped according to number of oocytes
Time Frame: On day of oocyte retrieval (up to 22 days after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Participants
  <4 Oocytes Retrieved | 13 | 26
  4-7 Oocytes Retrieved | 47 | 56
  8-14 Oocytes Retrieved | 84 | 82
  15-19 Oocytes Retrieved | 42 | 29
  >=20 Oocytes Retrieved | 16 | 11

6. Secondary Outcome: Number of Metaphase II Oocytes
Description: Only applicable for those inseminated using ICSI
Time Frame: On day of oocyte retrieval (up to 22 days after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: MII oocytes
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 96 | 99
MII oocytes | 9.2 (4.8) | 7.9 (4.7)
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Test type: Other; p = 0.0962, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = 1.11, 95% CI 2-sided [-0.20 to 2.41]

7. Secondary Outcome: Fertilization Rate
Description: Measured by the number of pronuclei. Fertilized oocytes with 2 pronuclei were regarded as correctly fertilized
Time Frame: On day 1 after oocyte retrieval (up to 23 days after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of fertilized oocytes
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 197 | 197
percentage of fertilized oocytes | 53.8 (24.1) | 54.4 (26.8)

8. Secondary Outcome: Number of Embryos
Description: The number of embryos (total and good-quality) was reported. Embryo quality is determined by combined assessment of cleavage stage (number of blastomeres/compaction status) and embryo morphology parameters
Time Frame: On day 3 after oocyte retrieval (up to 25 days after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Embryos
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Embryos
  Total number of embryos | 5.7 (3.9) | 5.0 (3.9)
  Number of good-quality embryos | 4.0 (3.2) | 3.9 (3.3)
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Number of embryos; Test type: Other; p = 0.1894, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = 0.51, 95% CI 2-sided [-0.25 to 1.27]
Statistical Analysis 2: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Number of Good-quality embryos; Test type: Other; p = 0.9361, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = -0.03, 95% CI 2-sided [-0.68 to 0.63]

9. Secondary Outcome: Number of Blastocysts
Description: The number of blastocysts (total and good-quality) was reported. Blastocyst quality is assessed by blastocyst expansion and hatching status, blastocyst inner cell mass grading, and trophectoderm grading. The scoring is based on the classification system by Gardner and Schoolcraft, with additional categories for inner cell mass (degenerative or no inner cell mass) and trophectoderm (degenerative or very large cells)
Time Frame: On day 5 after oocyte retrieval (up to 27 days after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Blastocysts
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Blastocysts
  Total Number of blastocysts | 3.8 (3.1) | 3.3 (2.9)
  Number of good-quality blastocysts | 2.3 (2.3) | 2.1 (2.2)
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Total number of blastocysts; Test type: Other; p = 0.2025, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = 0.37, 95% CI 2-sided [-0.20 to 0.94]
Statistical Analysis 2: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Number of good-quality blastocysts; Test type: Other; p = 0.5946, Negative binomial regression; Negative binomial regression model with treatment, age strata, and AMH group as factors; Difference = 0.12, 95% CI 2-sided [-0.31 to 0.54]

10. Secondary Outcome: Circulating Concentrations of Follicle-stimulating Hormone (FSH)
Description: Blood samples for analysis of circulating concentrations of FSH were drawn.
Time Frame: On stimulation day 6, at end-of-stimulation (up to 20 days after start of stimulation) and at oocyte retrieval (up to 22 days after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 199 | 200
IU/L
  Stimulation Day 6: number analyzed (Participants) | 198 | 198
  Stimulation Day 6 | 15.5 (4.3) | 16.7 (4.5)
  End-of-stimulation | 16.2 (4.4) | 15.8 (4.0)
  Oocyte retrieval: number analyzed (Participants) | 196 | 195
  Oocyte retrieval | 9.4 (2.8) | 9.8 (2.9)

11. Secondary Outcome: Circulating Concentrations of Luteinizing Hormone (LH)
Description: Blood samples for analysis of circulating concentrations of LH were drawn
Time Frame: as for outcome 10
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 199 | 200
IU/L
  Stimulation Day 6: number analyzed (Participants) | 199 | 198
  Stimulation Day 6 | 1.5 (0.9) | 5.6 (6.0)
  End-of-stimulation | 1.8 (0.9) | 1.8 (1.5)
  Oocyte retrieval: number analyzed (Participants) | 196 | 195
  Oocyte retrieval | 0.2 (0.2) | 2.0 (2.1)

12. Secondary Outcome: Circulating Concentrations of Estradiol
Description: Blood samples for analysis of circulating concentrations of estradiol were drawn
Time Frame: as for outcome 10
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 199 | 201
pmol/L
  Stimulation Day 6: number analyzed (Participants) | 198 | 200
  Stimulation Day 6 | 1190.1 (1101.2) | 2675.8 (1544.3)
  End-of-stimulation | 7542.7 (4106.8) | 6487.7 (3960.2)
  Oocyte retrieval: number analyzed (Participants) | 196 | 195
  Oocyte retrieval | 3485.1 (2129.0) | 3163.5 (1865.0)

13. Secondary Outcome: Circulating Concentrations of Progesterone
Description: Blood samples for analysis of circulating concentrations of progesterone were drawn
Time Frame: as for outcome 10
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 200 | 200
nmol/L
  Stimulation Day 6: number analyzed (Participants) | 198 | 198
  Stimulation Day 6 | 1.8 (1.0) | 2.6 (1.5)
  End-of-stimulation | 3.1 (1.4) | 3.5 (2.0)
  Oocyte retrieval: number analyzed (Participants) | 195 | 195
  Oocyte retrieval | 25.9 (12.9) | 26.0 (13.2)

14. Secondary Outcome: Circulating Concentrations of Inhibin B
Description: Blood samples for analysis of circulating concentrations of Inhibin B were drawn
Time Frame: as for outcome 10
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 196 | 198
pg/mL
  Stimulation Day 6: number analyzed (Participants) | 195 | 198
  Stimulation Day 6 | 690.4 (419.1) | 808.2 (428.5)
  End-of-stimulation: number analyzed (Participants) | 196 | 197
  End-of-stimulation | 1032.6 (605.2) | 938.1 (570.0)
  Oocyte retrieval: number analyzed (Participants) | 192 | 191
  Oocyte retrieval | 416.6 (253.9) | 389.0 (226.6)

15. Secondary Outcome: Total Gonadotropin Dose
Description: Calculated by start dates, end dates and daily dose of investigational medicinal product
Time Frame: Up to 20 days
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ug
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
ug | 112.2 (28.9) | 96.5 (26.0)
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Test type: Other; p < 0.0001, ANOVA; ANOVA model with treatment, age strata, and AMH group as factors; Difference = 16.94, 95% CI 2-sided [12.13 to 21.74]

16. Secondary Outcome: Number of Stimulation Days
Description: Calculated by start dates and end dates
Time Frame: Up to 20 days
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Days | 10.4 (1.9) | 8.8 (1.8)
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Test type: Other; p < 0.0001, ANOVA; ANOVA model with treatment, age strata, and AMH group as factors; Difference = 1.56, 95% CI 2-sided [1.19 to 1.92]

17. Secondary Outcome: Positive Beta Human Chorionic Gonadotropin (βhCG) Rate
Description: Defined as positive serum βhCG test
Time Frame: 13-15 days after transfer (up to approximately 1.5 months after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Participants
  Positive βhCG test | 91 | 79
  Negative βhCG test | 111 | 125
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Test type: Other; p = 0.1579, Regression, Logistic; Logistic regression model with treatment, age strata, and AMH group as factors; Difference = 6.99, 95% CI 2-sided [-2.71 to 16.70]

18. Secondary Outcome: Implantation Rate
Description: Defined as the number of gestational sacs after transfer divided by number of blastocysts transferred
Time Frame: 5-6 weeks after transfer (up to approximately 2.5 months after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Number; unit: Embryos
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 173 | 167
Embryos | 82 | 68

19. Secondary Outcome: Clinical Pregnancy Rate
Description: Defined as at least one gestational sac
Time Frame: 5-6 weeks after transfer (up to approximately 2.5 months after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Participants
  Positive | 81 | 68
  Negtaive | 121 | 136
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Test type: Other; p = 0.1134, Regression, Logistic; Logistic regression model with treatment, age strata, and AMH group as factors; Difference = 7.66, 95% CI 2-sided [-1.82 to 17.14]

20. Secondary Outcome: Vital Pregnancy Rate
Description: Defined as at least one intrauterine gestational sac with fetal heart beat
Time Frame: 5-6 weeks after transfer (up to approximately 2.5 months after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Participants
  Positive | 77 | 62
  Negative | 125 | 142
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Test type: Other; p = 0.0642, Regression, Logistic; Logistic regression model with treatment, age strata, and AMH group as factors; Difference = 8.81, 95% CI 2-sided [-0.52 to 18.14]

21. Secondary Outcome: Ongoing Pregnancy Rate
Description: At least one intrauterine viable fetus
Time Frame: 10-11 weeks after transfer (up to approximately 4 months after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Participants
  Positive | 73 | 60
  Negative | 129 | 144
Statistical Analysis 1: Comparison: FE 999049 + GnRH Agonist (GONAPEPTYL) vs FE 999049 + GnRH Antagonist (CETROTIDE); Test type: Other; p = 0.1002, Regression, Logistic; Logistic regression model with treatment, age strata, and AMH group as factors; Difference = 7.74, 95% CI 2-sided [-1.49 to 16.97]

22. Secondary Outcome: Ongoing Implantation Rate
Description: Defined as number of intrauterine viable fetuses divided by the number of blastocysts transferred
Time Frame: 10-11 weeks after transfer (up to approximately 4 months after start of stimulation)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Number; unit: Embryos
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 173 | 167
Embryos | 74 | 60

23. Secondary Outcome: Proportion of Subjects With Early OHSS (Including OHSS of Moderate/Severe Grade)
Description: Classification of grade was according to Golan's classification system, and all OHSS cases were graded as mild, moderate or severe.
Time Frame: Up to 9 days after triggering of final follicular maturation
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Participants | 8 | 5

24. Secondary Outcome: Proportion of Subjects With Late OHSS (Including OHSS of Moderate/Severe Grade)
Description: as for outcome 23
Time Frame: >9 days after triggering of final follicular maturation
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Participants | 4 | 6

25. Secondary Outcome: Frequency of Adverse Events
Description: Any untoward medical occurrence
Time Frame: From time of signing informed consent until the end-of-trial (approximately 7 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Participants | 112 | 109

26. Secondary Outcome: Intensity of Adverse Events
Description: Categorized as mild, moderate or severe
Time Frame: From time of signing informed consent until the end-of-trial (approximately 7 months)
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Percentage of participants
  Mild adverse events | 42.6 | 41.7
  Moderate adverse events | 18.8 | 16.7
  Severe adverse events | 4.0 | 3.4

27. Secondary Outcome: Technical Malfunctions of the Pre-filled Injection Pen
Description: Incidences of technical malfunctions of the pre-filled injection pen were recorded
Time Frame: Up to 20 days
Population: Participants analyzed for this endpoint represent participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
Number analyzed (Participants) | 202 | 204
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from signing of the informed consent until end-of-trial (approximately 7 months).
Description: Adverse events were recorded from signing of the informed consent until end-of-trial (approximately 7 months).
Arm/Group | FE 999049 + GnRH Agonist (GONAPEPTYL) | FE 999049 + GnRH Antagonist (CETROTIDE)
All-Cause Mortality (participants affected / at risk) | 0/202 | 0/204
Serious Adverse Events (participants affected / at risk) | 4/202 | 6/204
Other Adverse Events (participants affected / at risk) | 68/202 | 69/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 + GnRH Agonist (GONAPEPTYL) (N=202) | FE 999049 + GnRH Antagonist (CETROTIDE) (N=204)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 + GnRH Agonist (GONAPEPTYL) (N=202) | FE 999049 + GnRH Antagonist (CETROTIDE) (N=204)
Procedural pain (Injury, poisoning and procedural complications) | 20 (20) | 12 (12)
Headache (Nervous system disorders) | 27 (31) | 29 (30)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 10 (10) | 11 (11)
Pelvic pain (Reproductive system and breast disorders) | 14 (15) | 11 (12)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 12 (12) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT03809429/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT03809429/SAP_001.pdf